CLINICAL TRIAL: NCT05111327
Title: Skill Learning Abilities and Students' Self-confidence in Learning in High-fidelity Simulation: A Mixed Method
Brief Title: Skills Learning and Self-confidence in Learning in High-fidelity Simulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tung Wah College (Other)
Responsible Party: Principal Investigator, WONG Mei Fung Florence, Principal Investigator, Tung Wah College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: REC2021102
Record Dates: First submitted 2021-10-28; First posted 2021-11-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Problem-solving; Clinical Reasoning; Satisfaction
Keywords: Problem-solving, clinical reasoning, student satisfaction; clinical reasoning; student satisfaction; high-fidelity simulation; nursing education
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Students will be randomly assigned in either interventional group or control group. There are two facilitators. Each facilitator will be consistently responsible for either interventional group or control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The research assistant will assign students randomly in either interventional or control group. Students also did not know which group their facilitator is responsible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Students in the interventional groups will receive structured simulation guideline
  Interventions: Other: Structured guideline
- Control (No Intervention): Students in the control groups will receive standard treatment.

INTERVENTIONS:
Other: Structured guideline — Students in the intervention group will receive more learning materials before study. The structured guideline will be used to facilitate students' learning in simulation by the facilitator.
  Arms: Intervention

SUMMARY:
High-fidelity simulation (HFS) has become a favorable innovative teaching-learning method to facilitate students' learning in professional development in nursing. During the simulation, a variety of skills can be improved through HFS. This mixed randomized-control and qualitative study aims to examine the effects of the structured HFS guideline on PS, CR and Student Satisfaction and Self-Confidence in Learning in undergraduate nursing students and understand their learning experience in HFS.

DETAILED DESCRIPTION:
Nurses are facing new challenges of immediate clinical management for safer and higher quality of patient care in the current practice (Levette - Jones et al. 2018). Students are required to have independent learning and higher-intellectual skills, including problem-solving (PS) and clinical reasoning (CR), for pursuing better clinical judgements and decision-making and the most cost-effective practice (Levette - Jones et al. 2018). High-fidelity simulation (HFS) is one of the innovative and effective methods that allow students to apply integrated knowledge and skills in a designed simulated case scenario to develop higher-intellectual skills (Linn et al., 2012) and self-confidence. To allow students to achieve their HFS with enhancement of skill development and self-confidence in learning, a structured guideline is useful. This structured guideline can help course coordinators to maintain consistence in simulation teaching. Therefore, this study aims to understand students' skill development and self- confidence in learning through the HFS.

ELIGIBILITY:
Inclusion Criteria: Students who

* are undergraduate nursing students
* aged 18 or above

Exclusion Criteria: Students who

* are enrolled in the courses with high-fidelity simulation
* Have had clinical placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Problem-solving skills | 6 months
  Problem-solving Inventory (PSI) It consists of 32 items with a six-point Likert scale. The PSI includes three subscales: Problem-Solving Confidence (PSC) (11 items), Approach-Avoidance Style (AAS) (16 items) and Personal Control (PC) (5 items). PSC is to assess self-perceived confidence, belief and self-assurance effectively in solving problems. AAS is to measure an individual's tendency of response to approach or avoid problems. PC is to assess elements of self-control on emotions and behavior.
Nurses' Clinical Reasoning | 6 months
  Nurses' Clinical Reasoning Scale (NCRS) includes 15 items with a Likert five-point scale to assess students' CR competence. Higher scores indicate higher clinical reasoning competence.
Student Satisfaction and Self-Confidence in Learning | 6 months
  The Student Satisfaction and Self-Confidence in Learning consists of 13 items with 5-likert scales to measure students' perception of their satisfaction and self-confidence in learning. Five items are related to students' satisfaction in simulation-based learning activities and the remaining eight items concerns self-confidence in learning.

CONTACTS AND LOCATIONS:
Overall Officials: Florence MF Wong, Doctoral, Principal Investigator — Tung Wah College
Locations (1):
- Florence MF Wong, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
There is no plan to share IPD due to confidential data.
Supporting Information: ICF
Time Frame: June to August 2022
Access Criteria: Nurse educators Nurses Nurse students

REFERENCES:
- [Background] Cadorin L, Rei A, Dante A, Bulfone T, Viera G, Palese A. Enhancing self-directed learning among Italian nursing students: A pre- and post-intervention study. Nurse Educ Today. 2015 Jun;35(6):746-53. doi: 10.1016/j.nedt.2015.02.004. Epub 2015 Feb 18. PMID 25735910
- [Background] Heppner, P.P. & Petersen, C.H. The development and implications of a personal problem solving inventory. Journal of Counseling Psychology. 1982; 29: 66-75.
- [Background] Linn A, Khaw C, Kildea H, Tonkin A. Clinical reasoning - a guide to improving teaching and practice. Aust Fam Physician. 2012 Jan-Feb;41(1-2):18-20. PMID 22276278
- [Background] Liou SR, Liu HC, Tsai HM, Tsai YH, Lin YC, Chang CH, Cheng CY. The development and psychometric testing of a theory-based instrument to evaluate nurses' perception of clinical reasoning competence. J Adv Nurs. 2016 Mar;72(3):707-17. doi: 10.1111/jan.12831. Epub 2015 Oct 12. PMID 26455724
- [Background] Levett-Jones, T. (2nd Ed.). Clinical reasoning: Learning to think like a nurse. 2018. Pearson.
- [Background] National League for Nursing. Description of available tools. 2016. Retrieved from http://www.nln.org/professional-development-programs/research/tools-andinstruments/descriptions-of-available-instruments